CLINICAL TRIAL: NCT06248593
Title: Manually Controlled Continuous Infusion of Norepinephrine vs Phenylephrine During Spinal Anesthesia for Cesarean Section: A Double-blinded Randomized Controlled Study
Brief Title: Continuous Infusion of Norepinephrine vs Phenylephrine During Spinal Anesthesia for Cesarean Section (INPEACE)
Acronym: INPEACE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hassan II University (Other)
Responsible Party: Principal Investigator, Mohamed Adnane Berdai, Clinical professor, Hassan II University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EC01/2024
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Cesarean Section Complications; Hypotension
Keywords: hypotension; norepinephrine; cesarean delivery; Obstetric anesthesia; Spinal anesthesia; Phenylephrine
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Intervention Model Description: It's a randomized, double-blind, two-arm, parallel, non-inferiority, controlled trial, which tha aim is to test the hypothesis that neonatal outcome, as assessed by umbilical artery pH, is at least as good (non-inferior) when prophylactic continuous manually controlled infusion of norepinephrine is used to maintain blood pressure during spinal anaesthesia for elective cesarean delivery compared with the same infusion modalities of phenylephrine with more stable blood pressure and less bradycardia.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Before starting the study, a simple randomization sequence for at least 140 codes divided into two equal-sized groups will be generated. One code for each patient will be placed into a sealed, opaque, sequentially numbered envelope by a research assistant, who is not involved in patient management or data collection.
  A Medical staff member who is not involved in subsequent patient care or assessement either, will open the envelope for each patient shortly before commencement of the cesarean delivery and prepared two identical 50-mL syringes according to the code contained in the envelops, patients will be randomly allocated to receive Phenylephrine or Norepinephrine infusion. All the syringes will be labelled as "study drug", therefore it will be impossible for the anesthesiologists involved in patient care to identify whether it contained norepinephrine or phenylephrine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phenylephrine (Active Comparator): The infusion will have a concentration of Phenylephrine of 25 μg/mL and will be initiated at a rate of 96 mL/hour (1.6 mL/minute), that correspond to a phenylephrine rate infusion of 40 μg/min, then the infusion rate will be manually adjusted within the range 0-144 mL/h : PHE (0-60 μg/min).
  Interventions: Drug: Continuous infusion of Phenylephrine
- Norepinephrine (Experimental): The infusion will have a concentration of Norepinephrine of 4 μg/mL and will be initiated at a rate of 96 mL/hour (1.6 mL/minute), that correspond to norepinephrine rate infusion of 6.4 μg/min, then the infusion rate will be manually adjusted within the range 0-144 mL/h : Norepinephrine (0-9.6 µg/min).
  Interventions: Drug: Continuous infusion of Norepinephrine

INTERVENTIONS:
Drug: Continuous infusion of Norepinephrine — The rate of norepinephrine infusion will be adjusted according to values of systolic blood pressure measured noninvasively and recorded at 1-minute intervals along the intraoperative period, with the objective of maintaining values near baseline.
  Arms: Norepinephrine
Drug: Continuous infusion of Phenylephrine — The rate of phenylephrine infusion will be adjusted according to values of systolic blood pressure measured noninvasively and recorded at 1-minute intervals along the intraoperative period, with the objective of maintaining values near baseline.
  Arms: Phenylephrine

SUMMARY:
The goal of this clinical trial is to compare norepinephrine and ephedrine in maintaining blood pressure during spinal anaesthesia for elective cesarean delivery. The main questions it aims to answer are:

* Do phenylephrine and norepinephrine administered as manually controlled continuous infusion during elective cesarean delivery have different effects on neonatal outcome ?
* Do phenylephrine and norepinephrine administered as manually controlled continuous infusion during elective cesarean delivery have different effects on maternal hemodynamics? Participants will receive either phenylephrine or norepinephrine infusion, at the time of performing spinal anesthesia, the infusion rate will be adjusted manually depending on maternal arterial pressure.

DETAILED DESCRIPTION:
It's a randomized, double-blind, two-arm, parallel, non-inferiority, controlled trial that will be conducted in Hassan II University Hospital, Fes, Morocco. The aim of this study is to test the hypothesis that neonatal outcome, as assessed by potential of hydrogen (pH) of umbilical artery, is at least as good (non-inferior) when prophylactic continuous manually controlled infusion of norepinephrine (NE) is used to maintain blood pressure during spinal anaesthesia for elective cesarean delivery compared with the same infusion modalities of phenylephrine (PHE) with more stable blood pressure and less bradycardia.

Before starting the study, a simple randomization sequence will generate codes for two equal-sized groups. One code for each patient will be placed into a sealed, opaque, sequentially numbered envelope by a research assistant, who is not involved in patient management or data collection.

Another person not involved in subsequent patient care or assessement either, will open the envelope for each patient shortly before commencement of the study and prepared two identical 50-mL syringes according to the code contained in the envelops, patients will be randomly allocated to receive PHE or NE infusion. All the syringes were labelled as "study drug", To standardize and study the effects without affecting the potency of the drugs, vasopressor doses were taken in an equipotent ratio (12.5:1) for PHE:NE based on previous studies.

The medication used in this study are :

* NE : 4 ml vial of norepinephrine bitartrate injection, 2 mg/ml.
* PHE : 10 ml Phenylephrine hydrochloride pre-filled syringe 50 μg/ml. In group PHE, The infusion is prepared by taking 1 mg of phenylephrine (2 prefilled syringe equals to 20 ml) and diluting it with 0.9% normal saline (NS) to attain a total volume of 40 mL and a concentration of 25 μg/mL.

In group NE, Norepinephrine infusion will be prepared by taking one vial (8 mg) of norepinephrine, and diluting it with 496 ml of 0.9% normal saline (NS) to attain a concentration of NE of 16 µg/ml. 10 ml of this solution Will be diluted in 0.9% NS to reach a total volume of 40 mL and a concentration of 4 μg/mL of NE which correspond to 2 µg/ml of norepinephrine base.

Eleven milligrams of hyperbaric bupivacaine in addition to 20 μg fentanyl will be injected in the L2-L3, L3-L4 or L4-L5 intervertebral space using a 25-gauge pencil-point spinal needle in the sitting position. Block success will be assessed by sensory blockade level using pinprick test and surgery would not begin unless the sensory block reached T6 level. Patients with inadequate sensory blockade would receive general anesthesia for cesarean delivery, and will be excluded from the study.

Simultaneously with the intrathecal injection, rapid intravenous vascular volume expansion by 1000ml NS solution will be started, with a pressure infuser bag inflated.

The infusion will be initiated at a rate of 96 mL/hour (1.6 mL/minute), that correspond to a phenylephrine rate infusion of 40 μg/minute or norepinephrine rate infusion of 6.4 μg/minute. Both vasopressor infusions will be started at the same time that cerebrospinal fluid is obtained before the injection of the local anesthetic into the cerebrospinal fluid. and then manually adjusted within the range 0-144 mL/h : PHE (0-60 μg/min), NE (0-9.6 µg/min), according to values of systolic blood pressure (SBP) measured noninvasively and recorded at 1-minute intervals along the intraoperative period, with the objective of maintaining values near baseline, according to this modalities (table 1). Heart rate (HR) will be monitored continuously and recorded at 1-min interval.

SBP (% of baseline) Infusion rate (ml/min)) NE delivery rate (µg/min) PHE delivery rate (µg/min) >120% or >140 mmhg 0 0 0 100-120% 48 3.2 20 90-100% 96 6.4 40 80-90% 120 8 50 <80% 144 9.6 60

Table : Algorithm of manually controlled infusion rate and its corresponding amount of study drug (norepinephrine or phenylephrine depending on randomisation)

A researcher in the theater will manage the infusions and collect the data for analysis. Episodes of hypotension, hypertension, bradycardia and tachycardia will be recorded.

Intraoperative hypertension (defined as SBP greater than 120% of the baseline or > 140 mmhg) will be managed by stopping temporarily drug infusion. The infusion is resumed when blood pressure return to < 120% of the SBP baseline).

Postspinal hypotension (defined as decreased SBP less than 80% of the baseline or SBP< 90 mmhg reading during the period from intrathecal injection to delivery of the fetus) will be managed by increasing vasopressor infusion dose according to study protocol infusion above. In case of persistant postspinal hypotension despite increasing vasopressor doses, it's will be managed by 2-ml bolus of the infusion which correspond for parturients with NE infusion to 8µg and those with PHE to 50 μg. Additional vasopressor bolus will be given if SBP did not respond to the first dose within 2 min despite continuing the infusion.

In case of persistence of hypotension, A rescue bolus of at least ephedrine 6 mg is recommended, and repeated according to the severity and persistence of the hypotension.

After delivery and in the absence of hemorrhage, the vasopressor flow rate will be reduced in steps of 20 mL∙h-1, while maintaining an SBP >80% of baseline, a minimum delay of 5 minutes between 2 flow reductions is recommended to avoid secondary hypotension.

Intraoperative bradycardia (defined as heart rate less than 60 beats per minute without hypotension will be managed by stopping the vasopressor infusion.

If bradycardia is associated with hypotension, the patient will be managed by IV ephedrine 9 mg. If bradycardia persist or decrease below 50 beats/min after the previous measures, an IV atropine bolus (0.5 mg) should be given.

Umbilical arterial blood (UA) will be sampled from a double-clamped segment of umbilical cord by using arterial blood gas syringes. Within 20 min after clamping, umbilical blood gas will be analyzed with a bedside Blood gas Analyzer System.

ELIGIBILITY:
Inclusion Criteria:

* Full-term, singleton, pregnant women, nonlaboring.
* Scheduled for elective cesarean delivery under spinal anesthesia,
* American Society of Anesthesiologists physical status : 1 or 2
* Baseline systolic BP between 90 and 140 mm Hg.

Exclusion Criteria:

* Known fetal abnormality.
* Preexisting or pregnancy-induced hypertension, cardiovascular, cerebrovascular or kidney disease.
* Contraindication to spinal anesthesia.
* Peripartum hemorrhage.
* Body mass index above 40 kg/m2.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — As the study is about preventing hypotension in cesarean section. Only pregnant women are eligible.
Enrollment: 140 (Estimated)
Dates: Start 2025-01-29 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Umbilical artery pH | Immediately after delivery
  Umbilical arterial blood (UA) will be sampled from a double-clamped segment of umbilical cord by using arterial blood gas syringes.Umbilical blood gas will be analyzed with a bedside Blood gas Analyzer System.

SECONDARY OUTCOMES:
Umbilical artery base excess | Immediately after delivery
  From umbilical arterial blood gases.
Umbilical artery partial pressure of oxygen | Immediately after delivery
  From umbilical arterial blood gases.
Umbilical artery partial pressure of carbon dioxide | Immediately after delivery
  From umbilical arterial blood gases
APGAR score | 1 min after delivery
  A= Appearance P=Pulse G=Grimace A=Attitude R=Respiration. Values of APGAR score vary from 0 to 10, higher scores mean a better outcome.
APGAR score | 5 min after delivery
  A= Appearance P=Pulse G=Grimace A=Attitude R=Respiration. Values of APGAR score vary from 0 to 10, higher scores mean a better outcome.
Number of newborns admitted to neonatal intensive care unit | Within 24 hours after delivery
  Admission of the newborn to the neonatal intensive care unit
Blood glucose level from arterial umbilical cord blood gases | Immediately after delivery
  from arterial umbilical cord blood gases
Number of hypotensive episodes | from intrathecal injection to delivery of the fetus
  Defined as decreased systolic blood pressure intraoperatively less than 80% of the baseline or less than 90 mmhg
Number of severe hypotensive episodes. | from intrathecal injection to delivery of the fetus
  Defined as decreased systolic blood pressure intraoperatively less than 60% of the baseline or less than 70 mmhg
Number of episodes of bradycardia before delivery | From intrathecal injection to delivery of the fetus.
  Heart rate less than 60 beats per minute
Number of Hypertension episodes | In the intraoperative period.
  Systolic blood pressure at or above 120% of baseline
Number of episodes of Tachycardia | In the intraoperative period.
  Heart rate greater than 30% of baseline.
Number of episodes of nausea | From induction of spinal anesthesia to the end of the cesarean section.
  episodes of nausea experienced by patients
Number of episodes of vomiting | From induction of spinal anesthesia to the end of the cesarean section.
  Episodes of vomiting experienced by patients
Total dose of study drug given until delivery of the fetus. | From induction of spinal anesthesia to the delivery of the fetus
  The total dose given of norepinephrine or phenylephrine depending on randomization
Total dose of intraoperative study drug given. | From induction of spinal anesthesia to the end of the cesarean section.
  The total dose given of norepinephrine or phenylephrine depending on randomization
Total dose of ephedrine from induction of spinal anesthesia to delivery of the fetus. | from induction of spinal anesthesia to delivery of the fetus.
  Total dose of corrective boluses of ephedrine as a rescue drug
Total dose of intraoperative corrective boluses of ephedrine | From induction of spinal anesthesia to the end of the cesarean section.
  Total dose of corrective boluses of ephedrine as a rescue drug
Total dose of corrective boluses of atropine from induction of spinal anesthesia to delivery of the fetus. | from induction of spinal anesthesia to delivery of the fetus.
  Total dose of corrective boluses of atropine in case of bradycardia
Total dose of Intraoperative corrective boluses of atropine | From induction of spinal anesthesia to the end of the cesarean section.
  Total dose of corrective boluses of atropine in case of bradycardia

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Adnane Berdai, MD-PhD, Principal Investigator — University hospital Hassan II, Fes, Morocco
Locations (1):
- University hospital Hassan II, Fes, Morocco

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participant data will be shared and available to other researchers
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: the IPD and any additional supporting information will become available, 3 months after publication and will be available for a period of 6 months.
Access Criteria: Undecided now

REFERENCES:
- [Background] Heesen M, Stewart A, Fernando R. Vasopressors for the treatment of maternal hypotension following spinal anaesthesia for elective caesarean section: past, present and future. Anaesthesia. 2015 Mar;70(3):252-7. doi: 10.1111/anae.13007. Epub 2015 Jan 13. No abstract available. PMID 25583307
- [Background] Doherty DG, Norris S, Madrigal-Estebas L, McEntee G, Traynor O, Hegarty JE, O'Farrelly C. The human liver contains multiple populations of NK cells, T cells, and CD3+CD56+ natural T cells with distinct cytotoxic activities and Th1, Th2, and Th0 cytokine secretion patterns. J Immunol. 1999 Aug 15;163(4):2314-21. PMID 10438977
- [Background] Hasanin A, Aiyad A, Elsakka A, Kamel A, Fouad R, Osman M, Mokhtar A, Refaat S, Hassabelnaby Y. Leg elevation decreases the incidence of post-spinal hypotension in cesarean section: a randomized controlled trial. BMC Anesthesiol. 2017 Apr 24;17(1):60. doi: 10.1186/s12871-017-0349-8. PMID 28438121
- [Background] Veeser M, Hofmann T, Roth R, Klohr S, Rossaint R, Heesen M. Vasopressors for the management of hypotension after spinal anesthesia for elective caesarean section. Systematic review and cumulative meta-analysis. Acta Anaesthesiol Scand. 2012 Aug;56(7):810-6. doi: 10.1111/j.1399-6576.2011.02646.x. Epub 2012 Feb 7. PMID 22313496
- [Background] Stewart A, Fernando R, McDonald S, Hignett R, Jones T, Columb M. The dose-dependent effects of phenylephrine for elective cesarean delivery under spinal anesthesia. Anesth Analg. 2010 Nov;111(5):1230-7. doi: 10.1213/ANE.0b013e3181f2eae1. Epub 2010 Sep 14. PMID 20841418
- [Background] Ngan Kee WD, Lee SW, Ng FF, Tan PE, Khaw KS. Randomized double-blinded comparison of norepinephrine and phenylephrine for maintenance of blood pressure during spinal anesthesia for cesarean delivery. Anesthesiology. 2015 Apr;122(4):736-45. doi: 10.1097/ALN.0000000000000601. PMID 25635593
- [Background] Onwochei DN, Ngan Kee WD, Fung L, Downey K, Ye XY, Carvalho JCA. Norepinephrine Intermittent Intravenous Boluses to Prevent Hypotension During Spinal Anesthesia for Cesarean Delivery: A Sequential Allocation Dose-Finding Study. Anesth Analg. 2017 Jul;125(1):212-218. doi: 10.1213/ANE.0000000000001846. PMID 28248702
- [Background] Vallejo MC, Attaallah AF, Elzamzamy OM, Cifarelli DT, Phelps AL, Hobbs GR, Shapiro RE, Ranganathan P. An open-label randomized controlled clinical trial for comparison of continuous phenylephrine versus norepinephrine infusion in prevention of spinal hypotension during cesarean delivery. Int J Obstet Anesth. 2017 Feb;29:18-25. doi: 10.1016/j.ijoa.2016.08.005. Epub 2016 Aug 28. PMID 27720613
- [Background] Ngan Kee WD, Lee SWY, Ng FF, Khaw KS. Prophylactic Norepinephrine Infusion for Preventing Hypotension During Spinal Anesthesia for Cesarean Delivery. Anesth Analg. 2018 Jun;126(6):1989-1994. doi: 10.1213/ANE.0000000000002243. PMID 28678073
- [Background] Belin O, Casteres C, Alouini S, Le Pape M, Dupont A, Boulain T. Manually Controlled, Continuous Infusion of Phenylephrine or Norepinephrine for Maintenance of Blood Pressure and Cardiac Output During Spinal Anesthesia for Cesarean Delivery: A Double-Blinded Randomized Study. Anesth Analg. 2023 Mar 1;136(3):540-550. doi: 10.1213/ANE.0000000000006244. Epub 2022 Oct 24. PMID 36279409
- [Background] Ngan Kee WD. Phenylephrine infusions for maintaining blood pressure during spinal anesthesia for cesarean delivery: finding the shoe that fits. Anesth Analg. 2014 Mar;118(3):496-8. doi: 10.1213/ANE.0000000000000111. No abstract available. PMID 24557093
- [Background] Mohta M, Dubey M, Malhotra RK, Tyagi A. Comparison of the potency of phenylephrine and norepinephrine bolus doses used to treat post-spinal hypotension during elective caesarean section. Int J Obstet Anesth. 2019 May;38:25-31. doi: 10.1016/j.ijoa.2018.12.002. Epub 2018 Dec 13. PMID 30685301
- [Background] Ngan Kee WD. A Random-allocation Graded Dose-Response Study of Norepinephrine and Phenylephrine for Treating Hypotension during Spinal Anesthesia for Cesarean Delivery. Anesthesiology. 2017 Dec;127(6):934-941. doi: 10.1097/ALN.0000000000001880. PMID 28872480